CLINICAL TRIAL: NCT03936556
Title: A 3-Month Clinical Study to Assess the Effects of a Stannous Fluoride Dentifrice on Plaque and Gingivitis
Brief Title: A Clinical Study to Assess the Effects of a Stannous Fluoride Dentifrice on Plaque and Gingivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018004
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Marketed Stannous Fluoride Paste (Experimental): Brush twice daily
  Interventions: Drug: Marketed toothpaste
- Marketed Cavity Protection Toothpaste (Placebo Comparator): Brush twice daily
  Interventions: Drug: Marketed Cavity Protection Toothpaste

INTERVENTIONS:
Drug: Marketed toothpaste — Marketed stannous fluoride (0.454%) toothpaste
  Arms: Marketed Stannous Fluoride Paste
Drug: Marketed Cavity Protection Toothpaste — Marketed sodium monofluorophosphate (0.76 %) toothpaste
  Arms: Marketed Cavity Protection Toothpaste

SUMMARY:
The objective of this clinical study is to assess the effects of a 0.454% stannous fluoride dentifrice on gingivitis and plaque after 3 months when compared to a negative control.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent prior to participation and be given a signed copy of the informed consent form;
* Be in general good health as determined by the Investigator based on a review of the health history/update for participation in the trial;
* Have at least 16 gradable teeth;
* Agree to return for scheduled visits and follow the study procedures;
* Agree to refrain from use of any non-study oral hygiene products for the duration of the study;
* Agree to delay any elective dentistry, including dental prophylaxis, until the completion of the study;

Exclusion Criteria:

* Having taken antibiotic, anti-inflammatory, or anti-coagulant medications within 4 weeks of the Baseline Visit;
* Have any oral conditions that could interfere with study compliance and/or examination procedures, such as widespread caries, soft or hard tissue tumor of the oral cavity, or advanced periodontal disease;
* Removable oral appliances;
* Fixed facial or lingual orthodontic appliances;
* Self-reported pregnancy or lactation;
* Any diseases or condition that might interfere with the safe participation in the study; and
* Inability to undergo study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-02-25 (Actual); Primary Completion 2018-06-03 (Actual); Study Completion 2018-06-03 (Actual)

PRIMARY OUTCOMES:
Löe-Silness Gingivitis Evaluation | Baseline
  Löe-Silness Gingivitis Evaluation is a validated assessment of gingival health looking at inflammation and bleeding based on a 4 point range 0 (normal gingiva) to 3 (severe inflammation).
Löe-Silness Gingivitis Evaluation | 1 Month
  Löe-Silness Gingivitis Evaluation is a validated assessment of gingival health looking at inflammation and bleeding based on a 4 point range 0 (normal gingiva) to 3 (severe inflammation).
Löe-Silness Gingivitis Evaluation | 3 Months
  Löe-Silness Gingivitis Evaluation is a validated assessment of gingival health looking at inflammation and bleeding based on a 4 point range 0 (normal gingiva) to 3 (severe inflammation).

SECONDARY OUTCOMES:
Turesky Modified Quigley-Hein Index | Baseline
  The Turesky Modified Quigley-Hein Index is a validated assessment of dental plaque based on a scale of 0 (no plaque/debris) to 5 (plaque covering two-thirds or more of the side of the crown or tooth).
Turesky Modified Quigley-Hein Index | 1 Month
  The Turesky Modified Quigley-Hein Index is a validated assessment of dental plaque based on a scale of 0 (no plaque/debris) to 5 (plaque covering two-thirds or more of the side of the crown or tooth).
Turesky Modified Quigley-Hein Index | 3 Months
  The Turesky Modified Quigley-Hein Index is a validated assessment of dental plaque based on a scale of 0 (no plaque/debris) to 5 (plaque covering two-thirds or more of the side of the crown or tooth).

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Resources Group, Whittier, California, United States